CLINICAL TRIAL: NCT04055909
Title: Efficacy, Safety and Tolerability of Nangibotide in Patients With Septic Shock. A Randomized, Double-blind, Placebo Controlled Dose Selection Study
Brief Title: Efficacy, Safety and Tolerability of Nangibotide in Patients With Septic Shock
Acronym: ASTONISH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inotrem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOT-C-203; 2018-004827-36 (EudraCT Number)
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Shock, Septic
Keywords: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — nangibotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- nangibotide 1 (Experimental): Treatment with study drug at at dose of 0.3mg/kg/hr
  Interventions: Drug: nangibotide low dose
- nangibotide 2 (Experimental): Treatment with study drug at at dose of 1.0mg/kg/hr
  Interventions: Drug: nangibotide high dose
- Placebo (Placebo Comparator): Treatment with a matched placebo infusion
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: nangibotide low dose — nangibotide 0.3 mg/kg/h
  Other Names: LR12
  Arms: nangibotide 1
Drug: nangibotide high dose — nangibotide 1.0 mg/kg/h
  Other Names: LR12
  Arms: nangibotide 2
Drug: placebo — matching placebo
  Other Names: matched placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled dose-selection study in which two doses of nangibotide are tested versus placebo.

DETAILED DESCRIPTION:
All patients with a diagnosis of septic shock will be considered for study participation. All potential study patients will receive standard of care for the treatment of septic shock.

After screening for eligibility, patients meeting all inclusion and no exclusion criterion will be randomized. Patients will be randomized to one of three treatment arms.

Treatment with study drug must be initiated as early as possible, but no later than 24 hours after the onset of septic shock, defined by the start of vasopressor therapy.

Patients will be treated for at least 3 days with study drug. After the first 3 days of treatment, patients still requiring vasopressor will be treated until 24 hours after vasopressor withdrawal with a maximum treatment duration of 5 days.

Patients will be assessed at the End of Study (EoS) visit at day 28. After the last patient's day 28 visit, the study will be analyzed. Additional follow up (FU) visits will be conducted after 90 days, 6 and 12 months.

The objective of the study ist to compare the safety, tolerability and efficacy of two doses of nangibotide versus placebo, when given in addition to standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Age 18 to 85 years (inclusive)
3. Documented or suspected infection: lung, abdominal or urinary tract infection (UTI) in the elderly (≥65 years)
4. Organ dysfunction defined as acute change in total SOFA score ≥ 2 points
5. Refractory hypotension requiring vasopressors to maintain MAP ≥65mm Hg despite adequate volume resuscitation
6. Hyperlactatemia (blood lactate >2 mmol/L or 18 mg/dL).

Exclusion Criteria:

1. Previous episode of septic shock requiring vasopressor administration within current hospital stay
2. Underlying concurrent immunodepression with anti-CD52 alemtuzumab (Campath) or glucocorticoids >75 mg prednisone daily or equivalent for more than 7 days
3. Immunosuppressive therapy related to recent (<6 months) transplantation
4. Cancer chemotherapy (<3 months) implying an immunodepression
5. Known HIV infection with low CD4 cell count (<200) for at least 6 months
6. Known pregnancy (positive urine or serum pregnancy test)
7. Shock of any other cause, e.g. hypotension related to gastrointestinal bleeding
8. Ongoing documented or suspected endocarditis, history of prosthetic heart valves
9. Prolonged QT syndrome
10. End-stage neurological disease
11. End-stage cirrhosis (Child Pugh Class C)
12. Acute Physiology and Chronic Health Evaluation (APACHE II) score <15 or ≥ 34
13. Home oxygen therapy on a regular basis for > 6 h/day
14. Recent cardiopulmonary resuscitation (CPR) (within current hospital stay)
15. Body mass index (BMI) ≥ 40 kg/m2or weight ≥ 130 kg
16. Moribund patients
17. Decision to limit full care taken before obtaining informed consent
18. Participation in another interventional study in the 3 months prior to randomization

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2023-05-09 (Estimated)

PRIMARY OUTCOMES:
Sequential organ failure assessment (SOFA) score | day 5
  Change of total SOFA score from baseline to day 5 (in the subgroup defined by patients with elevated sTREM-1 baseline levels and in the overall population)

SECONDARY OUTCOMES:
All-cause mortality | day 5 and day 28
  all-cause mortality on D5 and D28
Duration of ICU stay | day 28
  hospitalization
Organe support free survival | day 28
  time to organe support free
Sepsis support index (SSI) | day 28
  Sepsis support index
Daily change of total Sequential organ failure assessment (SOFA) score and individual subscores | day 1, day 2, day 3, day 4, day 5, day 6 and day 7
  Daily change of total SOFA score and individual subscores
Duration of Vasopressor use | day 28
  Change in the Duration of Vasopressor use
Duration of Invasive mechanical ventilation (IMV) | day 28
  Change in the Duration of Invasive mechanical ventilation (IMV)
Duration of Renal support | day 28
  Change in the Duration of renal replacement therapy, RRT
All-cause mortality | 12 months
  all-cause mortality up to 12 months
Septic shock related mortality at day 28 | day 28
  mortality caused by septic shock
Incidence of secondary infections and post shock antibiotic use | day 28
  Incidence of secondary infections and post shock antibiotic use
Alive and organ support free at day 28 | day 28
  Proportion of patients alive and free of organ support at day 28
Overall survival on day 28 | day 28
  time from the date of study drug start to date of death from any cause
Overall survival up to 12 months | 12 months
  Overall survival up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Garaud, MD, Study Director — CEO and Medical Officer
Locations (43):
- Belgium (7):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Gent, Ghent
  - Centre hospitalier Jolimont-Lobbes, La Louvière
  - CHU Marie Curie, Lodelinsart
  - Clinique Saint-Pierre, Ottignies
  - CHU UCL Namur asbl, Yvoir
- Nordsjællandshospital Hillerød, Hillerød, Denmark
- Finland (3):
  - Helsinki University Hospital Adult ICU PPDS, Helsinki
  - Kuopion Yliopistollinen sairaala, Kuopio
  - Tampereen yliopistollinen sairaala, Tampere
- France (23):
  - CHU Angers, Angers
  - Centre hospitalier Victor Dupouy, Argenteuil
  - Centre hospitalier de Béthune, Béthune
  - Hôpital Fleyriat, Bourg-en-Bresse
  - CHU Dijon - Hôpital François Mitterrand, Dijon
  - CHD les Oudairies, La Roche-sur-Yon
  - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - CHU LE Mans, Le Mans
  - CHRU Lille - Hôpital Roger Salengro, Lille
  - Hôpital Universitaire Dupuytren, Limoges
  - Centre Hospitalier Lyon Sud, Lyon
  - Hôpital Nord, Marseille
  - Centre hospitalier de Melun, Melun
  - CHRU Nancy - Hôpital Central, Nancy
  - Hôtel Dieu - Nanates, Nantes
  - CHU de Nîmes, Nîmes
  - Hôpital de la source, Orléans
  - Hôpital Lariboisière, Paris
  - Hôpital Saint Louis, Paris
  - Groupe hospitalier Pitié-Salpêtrière, Paris
  - Hôpital Cochin, Paris
  - CHRU Hôpital Bretonneau, Tours
  - Hôpital d'instruction des Armées Robert Picqué, Villenave-d'Ornon
- Ireland (2):
  - St Jame's Hospital, Dublin
  - Galway University Hospital, Galway
- Spain (7):
  - Hospital del mar, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Clinical San Carlos, Madrid
  - Hospital Universitario Dentral de Asturias, Oviedo
  - Hospital Universitari Mutua de Terrassa, Terrassa
  - Hospital universitario DR. Peset Aleixandre, Valencia
  - Hospital Universitario y Politecnico la Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Francois B, Lambden S, Fivez T, Gibot S, Derive M, Grouin JM, Salcedo-Magguilli M, Lemarie J, De Schryver N, Jalkanen V, Hicheur T, Garaud JJ, Cuvier V, Ferrer R, Bestle M, Pettila V, Mira JP, Bouisse C, Mercier E, Vermassen J, Huberlant V, Vinatier I, Anguel N, Levy M, Laterre PF; ASTONISH investigators. Prospective evaluation of the efficacy, safety, and optimal biomarker enrichment strategy for nangibotide, a TREM-1 inhibitor, in patients with septic shock (ASTONISH): a double-blind, randomised, controlled, phase 2b trial. Lancet Respir Med. 2023 Oct;11(10):894-904. doi: 10.1016/S2213-2600(23)00158-3. Epub 2023 May 31. PMID 37269870
- [Derived] Francois B, Lambden S, Gibot S, Derive M, Olivier A, Cuvier V, Witte S, Grouin JM, Garaud JJ, Salcedo-Magguilli M, Levy M, Laterre PF. Rationale and protocol for the efficacy, safety and tolerability of nangibotide in patients with septic shock (ASTONISH) phase IIb randomised controlled trial. BMJ Open. 2021 Jul 7;11(7):e042921. doi: 10.1136/bmjopen-2020-042921. PMID 34233965